CLINICAL TRIAL: NCT00718276
Title: Pharmacokinetic Study in Healthy Postmenopausal Women to Compare Supplementation of Vitamin D3 to 25(OH)D
Brief Title: Pharmacokinetic Study: Effect of 25(OH)D and Vitamin D3 on Serum 25(OH)D
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007-09-13-HyD
Record Dates: First submitted 2008-07-17; First posted 2008-07-18 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: Healthy postmenopausal women
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 25(OH)D
  Interventions: Drug: 25(OH)D
- 2 (Active Comparator): vitamin D3
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Drug: 25(OH)D — daily (20ug), weekly (140 ug), Bolus (140 ug)
  Other Names: HyD
  Arms: 1
Dietary Supplement: vitamin D3 — daily (800 IU), weekly (5600 IU), Bolus (5600 Iu)
  Other Names: Cholecalciferol
  Arms: 2

SUMMARY:
We compare the effect of HyD (25-hydroxyvitamin D) and vitamin D3 in their effect on 25-hydroxyvitamin D plasma levels over a course of 4 month. This is a pharmacokinetic study including 35 postmenopausal women.

* Trial with medicinal product

DETAILED DESCRIPTION:
We include postmenopausal women age 50 to 75, race/ethnicity: Caucasian, serum 25(OH)D at baseline between 20 to 60 nmol/l, body mass index: < 30 kg/m2

to compare 25(OH)D and vitamin D3 in equimolar doses over a 4 month pharmacokinetic trial. The dosing arms are daily, weekly, and bolus

ELIGIBILITY:
Inclusion criteria:

* Postmenopausal women
* Age 50 to 75 years
* Body mass index 18-29 kg/m2
* 25-hydroxyvitamin D levels 20 to 60 nmol/l
* Caucasian
* Generally healthy

Exclusion criteria:

* Serum calcium > 2.6 nmol/L
* Use if dietary supplements (> 400 IU vitamin D per day, > 600 mg of calcium per day)
* Hypertension
* Diseases that carry the risk of hypercalcemia
* Use of any drug that interferes with bone metabolism in the last 12 months (bisphosphonates estrogen receptor modulators, PTH, calcitonin)
* Oral HRT in the last 6 months
* Extreme diets
* Fracture or fall in the last 3 months
* Current smoking or alcohol abuse
* Planning on a sunny vacation in the course of the trial
* Kidney stone history
* Creatinine clearance < 30 ml/min
* Co-medications: anticoagulants, PTH, corticosteroids, thiazide diuretics, digoxin, anticonvulsants, malabsorption,z C

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-03; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
serum 25(OH)D levels | repeated assessments over 4 months

SECONDARY OUTCOMES:
muscle strength, blood pressure, blood glucose, bone markers | repeated assessments over 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Heike Bischoff Ferrari, MD, MPH, Principal Investigator — University Hospital Zurich, Centre on Aging and Mobility
Locations (1):
- University Hospital Zurich, Centre on Aging and Mobility, Zurich, Canton of Zurich, Switzerland